CLINICAL TRIAL: NCT06631781
Title: Cognitive Control Amongst Older Adults with Depressive Symptom: Mechanisms and Intervention
Brief Title: Cognitive Control Mechanisms in Older Adults
Acronym: GOLD-Cog+
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hebrew University of Jerusalem (Other)
Collaborators: University of Melbourne (Other)
Responsible Party: Principal Investigator, Mor Nahum, Professor, Hebrew University of Jerusalem
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: GOLD-Cog+
Record Dates: First submitted 2024-06-30; First posted 2024-10-08 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-06

CONDITIONS: Depressive Symptoms
MeSH Terms: conditions — Depression

STUDY DESIGN:
Intervention Model Description: Participants will participate in both a 6-week experimental period and a 6-week waiting period
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- GOLD-Cog+ (Experimental): The experimental group receives 6 weeks of combined cognitive intervention (GOLD-Cog+),which includes participation in 9, one hour long Cognitive-Orientation to Occupational Performance(CO-OP)-based group sessions and 24 individual and independent 30-minute computerized cognitive training (CCT) program using the Effectivate platform (Israeli-based CCT developed for older adults. Available in both Hebrew and English).
  Interventions: Other: GOLD-Cog+
- Waiting period (No Intervention): The same participants will also participate in 6-weeks of no intervention before or after the 6-week experimental period (i.e. crossover study). This will be used as the 'control' group.

INTERVENTIONS:
Other: GOLD-Cog+ — 6 weeks of combined cognitive intervention (GOLD-Cog+),which includes participation in 9, one hour long Cognitive-Orientation to Occupational Performance(CO-OP)-based group sessions and 24 individual and independent 30-minute computerized cognitive training (CCT) program using the Effectivate platform (Israeli-based CCT developed for older adults. Available in both Hebrew and English).
  Other Names: CCT + functional-based approach (CO-OP)
  Arms: GOLD-Cog+

SUMMARY:
The prevalence of depressive symptoms in older adults is on the rise, affecting 13 to 37% of older adults globally. These symptoms significantly impact health, increasing the risk of dementia and cognitive decline, and impairing daily functioning and quality of life. Reduced cognitive control (CC) is a key factor contributing to depressive symptoms, affecting 40% of adults with such symptoms. Despite this, over half of affected adults do not respond well to available treatments. Computerized cognitive training (CCT) has shown efficacy in improving CC but its impact on daily functioning is limited. The Cognitive Orientation to Occupational Performance (CO-OP) approach has demonstrated promise in improving daily functioning, as measured by occupational performance (OP). We propose a novel intervention, GOLD-Cog+, combining CCT and CO-OP, to address CC and functional deficits in older adults with depressive symptoms.

DETAILED DESCRIPTION:
The goal of this clinical trial is to investigate the relationship between mood and cognitive control in community-dwelling older adults (65+) with sub-clinical depression and to assess feasibility, efficacy, and sustainability of a proposed combined cognitive intervention, GOLD-Cog+, for this population group. Cognitive control is the mental abilities that underlie our goal-directed behavior. These mental abilities include: the ability to shift our attention, constantly monitoring and updating information provided by our environment and having the ability to inhibit unwanted reactions.

The main questions of this study are:

Question 1: What is the relationship between mood and cognitive control in daily life of older adults with depressive symptoms? Question 2: Can this proposed combined cognitive intervention, GOLD-Cog+ help improve daily functioning, cognitive control, mood, quality of life and subjective cognition in older adults with depressive symptoms? Question 3: Are the participants satisfied with this new proposed intervention?

Participants will participate in a crossover randomized control trial in which they will participate in a 6-week experimental period and a 6-week waiting period. During the experimental period, they will take part in individual computerized cognitive training and functional-based, goal-oriented group sessions.

ELIGIBILITY:
Inclusion Criteria:

* Depressive Symptoms based on Patient Health Questionnaire (PHQ-8) ≥ 5
* Healthy Cognition based on Montreal Cognitive Assessment (MoCa) ≥ 20
* Capable of signing and agreeing to participate in the study
* Have the basic technological skills to use a tablet based on self-report
* Adequate sight and hearing abilities (with assistive technology) to be able to use a tablet and fully participate in a small group setting (6 people)
* Ability to fluently read, speak and understand Hebrew or English

Exclusion Criteria:

* Any neurodegenerative disorder (e.g., Mild Cognitive Impairment (MCI), Dementia, Parkinson's disease) via self-report
* Psychiatric disorders, not including depression or anxiety disorders (specifically: Schizophrenia, Bipolar or Psychotic disorders) via self-report

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2024-02-02 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Adaptive Cognitive Evaluation (ACE) Battery | Pre-test, post-test (7-weeks after pre-test)
  An online assessment tool, comprised of 6 sub-tasks based on standardized tests to assess cognitive control (inhibition, shifting, monitoring) in an immersive and user-friendly interface
Canadian Occupational Performance Measure (COPM) | Pre-test, post-test (7-weeks after pre-test)
  Used to measure functioning by measuring occupational performance. The COPM is a semi-structured interview rating clients' self-perception of performance and satisfaction in their five most important functional problems. Importance, performance, and satisfaction for each goal are rated on a 10-point Likert scale, with 1 denoting not important at all, not satisfied at all and not able to do it at all, and 10 denoting extremely important, able to do it extremely well and extremely satisfied, respective of the scale used

SECONDARY OUTCOMES:
Beck Depression Scale (BDI-II) | Pre-test, post-test (7-weeks after pre-test)
  Used to measure depressive symptomsThe BDI-II is a 21-item, self-administered questionnaire which requires 5-to-10-minutes to complete, aimed at measuring the severity of depression in diagnosed patients, as well as detecting possible depression in the normal population above the age of 13. Each question refers to the previous 2 weeks and is rated on a 4-point Likert scale, with scores ranging from 0 (absence of a given symptom) to 3 (maximum level of severity). Total scores range between 0-63 where a higher score indicates a higher severity of depression .
State Trait Anxiety Inventory (STAI) tool | Pre-test, post-test (7-weeks after pre-test)
  Used to measure anxiety. It is a 20-item self-administered questionnaire regarding one's general feelings of anxiety at the present moment, using a 4-point Likert scale, with scores ranging from 1 (not at all) to 4 (very). Total scores range between 4-80 where a higher score indicates a higher level of anxiety.
The Older People's Quality of Life (OPQoL-35) | Pre-test, post-test (7-weeks after pre-test)
  Used to measure quality of life. It is a 35-item self-administered questionnaire designed to capture the older adult's quality of life needs. Each question is scored on a 5-point Likert Scale, from 1 (strongly agree) to 5 (do not agree at all). Total scores range from 35 to 175, where a higher score indicates better quality of life.

OTHER OUTCOMES:
Cognitive Orientation to Occupational Performance (CO-OP) fidelity checklist | Post-intervention (7-weeks after pre-test)
  Used to ensure a high standard of procedural fidelity of the CO-OP intervention,
Ruminative Response Scale (RRS-22) | Pre-test, post-test (7-weeks after pre-test), follow-up (14 weeks after pre-test)
  Used to measure trait rumination. It is a 22-item, self-administered questionnaire regarding one's general way of thinking, using a 4-point Likert scale, from 1 (almost never) to 4 (almost always) with total scores range from 4-88, where a higher score indicates a higher level of rumination
Performance Quality Rating Scale (PQRS) | Pre-test, post-test (7-weeks after pre-test), follow-up (14 weeks after pre-test)
  a 10-point scale used to measure daily functioning, by measuring occupational performance of client-selected activities. 1 means poor performance, with 10 meaning excellent performance
Intrinsic Motivation Inventory (IMI) | Post-intervention (7-weeks after pre-test)
  used to measure participants' subjective experience of their participation in the study
Cognitive Failures Questionnaire (CFQ) | Pre-test, post-test (7-weeks after pre-test), follow-up (14 weeks after pre-test)
  Used to measure subjective cognition. The CFQ will be used to measure subjective cognition. It is a 25-item questionnaire, with a scale of 0 to 4, where 4 is very often and 0 is never. Total score is out of 100.
Satisfaction questionnaire and a semi-structured interview | Post-intervention (7-weeks after pre-test)
  Used to measure the participants' satisfaction with the study, specifically regarding the group meetings

CONTACTS AND LOCATIONS:
Locations (1):
- Computerized Neurotherapy Lab, School of OT, Hebrew University, Mt. Scopus Campus, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: No